CLINICAL TRIAL: NCT01284738
Title: Beta-thalassemia and Microparticles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010-A00198-31; 2009-18
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Thalassemia Major (TM); Thalassemia Intermedia (TI); Microparticles (MP)Originating From Platelets, Endothelial Cells and Monocytes
Keywords: TM; TI; MP
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TM patients (Active Comparator): thalassemia major (TM) Need transfusion for survive
  Interventions: Other: Physiopathology
- TI patients (Active Comparator): thalassemia intermedia (TI) Patients with TI have a milder clinical phenotype than those with TM
  Interventions: Other: Physiopathology

INTERVENTIONS:
Other: Physiopathology — Three sequential biological evaluations will be performed for each patient and will consist in :
  * the dosages of MP carried out by the UMR 608 in Marseille,
  * the evaluation of the oxidative stress markers and of iron performed in the UMR 773 in Paris-Bichat.
  In vitro production of MP of transfused red blood cells origin will also be evaluated in erythrocytes concentrates during the storage of the units.
  Arms: TM patients
Other: Physiopathology — Three sequential biological evaluations will be performed for each patient and will consist in :
  * the dosages of MP carried out by the UMR 608 in Marseille,
  * the evaluation of the oxidative stress markers and of iron performed in the UMR 773 in Paris-Bichat.
  Arms: TI patients

SUMMARY:
The results will allow us to evaluate the role of MP in the thrombo-embolic risk observed in thalassemic patients and to underline a possible difference between TM and TI. The in vitro and in vivo study of MP in erythrocytes concentrates is a new approach to explore the consequence of transfusion in polytransfused patients. Finally, the identification of a possible relationship between the oxidative stress and the production of MP may lead to the development of specific therapeutical approaches

DETAILED DESCRIPTION:
Microparticles (MP) are intact vesicles derived from cell membranes which arise mainly through cell membrane activation processes and from apoptosis. MP originating from platelets, endothelial cells and monocytes have been most extensively studied, though similar particles can arise from red cells and granulocytes. The ability to form microparticles is an essential part of physiological coagulation.However, MP may play an important procoagulant role in several diseases including sickle cell disease, and paroxysmal nocturnal haemoglobinuria (PNH).

Several studies reported the presence of MP in TI and their potential role in the hypercoagulable state. The investigators propose in this study to investigate the presence and origin of MP in TM patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient recorded in the national register of the patients attained by beta-thalassemia (TI) or (TM)
* Patient monitoring in one of 5 recruiters centers
* Patient more than 15 years
* Patient consented and informed

Exclusion Criteria:

* Blood transfusion dating from less than 3 months for TI
* Composite Heterozygotes HbE /beta-thalassemia
* pregnant women
* other disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Relationship between TM and TI | 36 months
  * In TM, to quantify the elevation of MP as well as their procoagulant activity, to describe their production kinetic, to determine the transfusional or endogenous origin of erythrocytic MP and finally to compare their characteristics with those found in TI patients.
  * To study, in TM and TI patients, the relationship between the number, the procoagulant activity of MP and the clinical (thromboembolic episodes,splenectomy, presence of pulmonary hypertension) biological and plasmatic data reflecting the patient's prothrombotic state.

SECONDARY OUTCOMES:
Investigate the mechanisms of the elevated production of MP in thalassemias | 36 months
  Studying the correlation between the number, the activity of erythrocytes and platelets derived-MP and the hemolysis, the dyserythropoiesis, the oxidative stress and iron overload markers.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Thuret, Doctor, Study Director — APHM
Locations (1):
- APHM, Marseille, France